CLINICAL TRIAL: NCT06417476
Title: A Multicenter, Open, Randomized, Phase II Trial：Short-course Radiotherapy or Long-course Chemoradiation Followed by MFOLFOXIRI Consolidation Chemotherapy for Organ Preservation in Low Rectal Cancer
Brief Title: Short-course Radiotherapy or Long-course Chemoradiation Followed by MFOLFOXIRI Consolidation Chemotherapy for Organ Preservation in Low Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pei-Rong Ding (Other)
Collaborators: Yunnan Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Shantou Central Hospital (Other); Fujian Cancer Hospital (Other Government); Jiangsu Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Pei-Rong Ding, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-714
Record Dates: First submitted 2024-02-04; First posted 2024-05-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-05

CONDITIONS: Rectal Neoplasms
Keywords: Neoadjuvant chemotherapy; Preoperative radiotherapy; Chemoradiotherapy; Consolidation chemotherapy; mFOLFOXIRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — Irinotecan; Oxaliplatin; formic acid; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short-course radiotherapy followed by consolidation chemotherapy with mFOLFOXIRI (Experimental): Patients receive short-course radiotherapy (25Gy/5 times) followed by consolidation chemotherapy with mFOLFOXIRI (Irinotecan 150 mg/m2 iv gtt (2h) d1, Oxaliplatin 85 mg/m2 iv gtt (2h) d1, Calcium folinate 400 mg/m2 iv gtt (2h) d1, Total amount of fluorouracil 2400 mg/m2 iv gtt (48h)), treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. The first efficacy evaluation occurs after the fourth chemotherapy cycle. If there is no progression (a complete response (CR), partial response (PR), or stable disease (SD) with reduction or stability in tumor size) , patients will proceed with an additional four cycles. Upon the final efficacy assessment after the eighth chemotherapy cycle, patients will received several pathways (watch & wait approach; local resection;total mesorectal excision) are considered based on the assessments.
  Interventions: Radiation: Short-course radiotherapy; Drug: Irinotecan; Drug: Oxaliplatin; Drug: Calcium Formate; Drug: Fluorouracil
- Long-course chemoradiation followed by consolidation chemotherapy with mFOLFOXIRI (Experimental): Patients receive long-course chemoradiation (50Gy/25 times;capecitabine 825 mg/m² twice daily) followed by consolidation chemotherapy with mFOLFOXIRI (Irinotecan 150 mg/m2 iv gtt (2h) d1, Oxaliplatin 85 mg/m2 iv gtt (2h) d1, Calcium folinate 400 mg/m2 iv gtt (2h) d1, Total amount of fluorouracil 2400 mg/m2 iv gtt (48h)), treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. The first efficacy evaluation occurs after the fourth chemotherapy cycle. If there is no progression (a complete response (CR), partial response (PR), or stable disease (SD) with reduction or stability in tumor size) , patients will proceed with an additional four cycles. Upon the final efficacy assessment after the eighth chemotherapy cycle, patients will received several pathways (watch & wait approach; local resection;total mesorectal excision) are considered based on the assessments.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Calcium Formate; Drug: Fluorouracil; Radiation: Long-course chemoradiation; Drug: Capecitabine

INTERVENTIONS:
Radiation: Short-course radiotherapy — The total dosage was 25Gy consisted of 5 fractions of 5 Gy to clinical target volume without a boost dose
  Arms: Short-course radiotherapy followed by consolidation chemotherapy with mFOLFOXIRI
Drug: Irinotecan — 150 mg/m² iv drip over 2 hours on day 1, repeated every 14 days.
Drug: Oxaliplatin — 85 mg/m² iv drip over 2 hours on day 1, repeated every 14 days.
Drug: Calcium Formate — 400 mg/m² iv drip over 2 hours on day 1, repeated every 14 days.
Drug: Fluorouracil — 2400 mg/m² iv drip over 48 hours on day 1-2, repeated every 14 days.
Radiation: Long-course chemoradiation — The total dosage was 50Gy consisted of 25 fractions of 2 Gy to clinical target volume without a boost dose
  Arms: Long-course chemoradiation followed by consolidation chemotherapy with mFOLFOXIRI
Drug: Capecitabine — 825 mg/m² twice daily administered orally and concurrently with radiation therapy for 5 days per week.
  Arms: Long-course chemoradiation followed by consolidation chemotherapy with mFOLFOXIRI

SUMMARY:
Given the growing focus on preserving organ function and the utilization of neoadjuvant therapy, it is important to investigate and enhance the application of comprehensive neoadjuvant therapy in low rectal cancer. This approach aims to minimize or circumvent the organ dysfunction and subsequent decline in quality of life associated with radical surgery, with improving disease-free survival (DFS), while . Consequently, we propose to initiate a multicenter clinical trial to examine the medium- and long-term effectiveness of complete neoadjuvant therapy (comprising either short-course radiotherapy or long-course chemoradiation, followed by consolidation chemotherapy with mFOLFOXIRI) in increasing organ preservation rates in patients with low rectal cancer.

DETAILED DESCRIPTION:
This randomised, open-label, multicentre,phase II trial began in December, 2022, as a neoadjuvant trial about short-course radiotherapy or long-course chemoradiation followed by mFOLFOXIRI consolidation chemotherapy,in patients aged 18 years to 70 with clinical stage II-III locally advanced low rectal cancer from six Chinese institutions. The primary endpoint of the study was the 1-year organ preservation rate, with a comparison to historical data. Additionally, the study compared the differences between two radiotherapy regimens within the TNT treatment and explored biomarkers to predict tumor response

Patients with local advanced rectal cancer (cT2-4aN0-2,M0, 8cm from the anus verge) were recruited. Patients receive short-course radiotherapy (25Gy/5 times) followed by consolidation chemotherapy or long-course chemoradiation (50Gy/25 times;capecitabine 825 mg/m² twice daily) with mFOLFOXIRI (Irinotecan 150 mg/m2 iv gtt (2h) d1, Oxaliplatin 85 mg/m2 iv gtt (2h) d1, Calcium folinate 400 mg/m2 iv gtt (2h) d1, Total amount of fluorouracil 2400 mg/m2 iv gtt (48h)), treatment repeats every 14 days for 8 courses in the absence of disease progression or unacceptable toxicity. The efficacy evaluation occurs after the fourth and eighth chemotherapy cycle. Patients showing a complete response (CR), partial response (PR), or stable disease (SD) with reduction or stability in tumor size are advised to continue and complete all planned consolidation chemotherapy. However, if the evaluation indicates stable disease with an increase (SD increased) or progressive disease (PD), and if an R0 resection (complete removal of the tumor with no cancer cells at the margins) is feasible, radical total mesorectal excision (TME) should be pursued. In cases where R0 resection is not achievable, the treatment should align with the guidelines for managing unresectable rectal cancer. Upon the final efficacy assessment after the eighth chemotherapy cycle, several pathways are considered based on the outcomes: patients achieving a clinical complete response (cCR) may proceed to a Watch & Wait approach. Those with a near clinical complete response (near cCR) undergo local transanal resection. If the patient's condition is evaluated as PR/SD with a reduction but does not qualify as near cCR, radical TME is recommended. For patients showing SD with an increase or PD, yet with a potential for R0 resection, radical TME is again the suggested course of action. If R0 resection is unattainable, treatment should adhere to the guidelines for unresectable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: Histologically confirmed rectal adenocarcinoma. Preoperative Staging: Clinical stages cT2-4aN0-2. Tumor Location: Tumor's lower edge within 8cm from the anus, potentially affecting anal preservation or function.

Metastasis Screening: Preoperative chest, abdomen, and pelvis CT to rule out distant metastasis.

Biomarkers: Positive expression of pMMR (MSH1/MSH2/MSH6/PMS2) on tumor biopsy immunohistochemistry.

Staging Methods: Combination of thoracic and abdominal pelvic CT, pelvic MRI, and endoscopic or transrectal ultrasound.

Patient Characteristics Age: 18 to 70 years. Performance Status: ECOG score of 0-1. Life Expectancy: At least 2 years. Blood Counts: WBC >4000/mm^3, PLT >100,000/mm^3, Hb >10g/dL (chronic anemia with Hb < 10.0g/dL subject to multidisciplinary team review).

Liver Function: Serum total bilirubin ≤1.5×ULN (≤3×ULN for Gilbert syndrome); AST and ALT ≤2.5×ULN.

Renal Function: Serum creatinine ≤1.5×ULN or creatinine clearance >50 mL/min. Other Criteria: Non-pregnant, not nursing, no other malignancies (except non-melanoma skin cancer or cervical carcinoma in situ) within the past 5 years, capable of providing informed consent, no severe comorbidities affecting survival.

Prior Treatment No prior surgery, chemotherapy, or radiotherapy for rectal cancer. No prior biological therapy. No restrictions on previous endocrine therapy.

Exclusion Criteria:

Informed Consent: Lack of signed informed consent. Genetic Markers: Tumor biopsy indicating dMMR or MSI-H detected. Advanced Tumor Stage: Preoperative assessment showing tumor invasion of surrounding tissues/organs (T4b).

Obstruction: Unresolved colonic obstruction; presence of tumor perforation. Metastasis: Evidence of preoperative distant metastasis. Cardiac Conditions: Arrhythmia requiring antiarrhythmic therapy (excluding beta-blockers or digoxin), symptomatic coronary artery disease or recent myocardial ischemia (within 6 months), or congestive heart failure above NYHA Grade II.

Hypertension: Severe, poorly controlled hypertension. Infections: HIV infection, active chronic hepatitis B or C, other serious infections; active tuberculosis or anti-TB therapy within the past year.

Organ Function: Poor fluid quality, organ function decompensation. Previous Treatment: History of pelvic or abdominal radiotherapy; multiple primary colorectal cancers.

Neurological Conditions: Seizures requiring management (e.g., steroids, antiepileptic therapy).

Cancer History: Other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ or basal cell carcinoma of the skin.

Substance Abuse: Substance abuse or medical, psychological, or social conditions affecting study participation or result evaluation.

Allergies: Known or suspected allergy to study drugs or related medications. Stability: Any unstable condition that may compromise safety or compliance. Reproductive Status: Pregnant or lactating women, or fertile women not using effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate | Up to 1 years
  The 1-year organ preservation rate is the percentage of patients attaining a complete clinical response (cCR) or near-complete clinical response (near-cCR) following neoadjuvant therapy, who then proceeded with non-surgical management or local excision, was monitored under a Watch & Wait strategy or for 1 year post-local resection without undergoing radical surgery.

SECONDARY OUTCOMES:
Clinical complete response | Up to 24 weeks
  The definition of a cCR is (1) substantial downsizing with no residual tumor or residual fibrosis only (with low signal on high b-value DWI, if available), shown in Figure 1. Residual wall thickening due to edema only was also an indication for a possible cCR ; (2) no suspicious lymph nodesonMRI; (3) no residual tumor at endoscopyor onlya small residual erythematousulcer or scar; (4) negative biopsiesfromthe scar, ulcer, orformertumorlocation;and (5)nopalpabletumor,wheninitially palpable with digital rectal examination
Pathological complete response | Up to 24 weeks
  Pathological response will be made based on assessment of the surgical specimen at the primary treatment site. This assessment is made in addition to the AJCC 7th edition summary staging. A pCR must include no gross or microscopic tumor identified anywhere within the surgical specimen. This must include:
  No evidence of malignant cells in the primary tumor specimen No lymph nodes that contain tumor. The definition of a non-pCR will include any surgical specimen that has any evidence of residual tumor manifest in the primary or regional lymph nodes. For patients who do not meet criteria for a pCR, the extent of response to preoperative therapy will be graded using the Tumor Regression Grade (TRG) schema that is included in the AJCC 7th edition. This was also used by Rodel in the pre/postoperative rectal cancer study and was subsequently adopted by the AJCC [Rodel (JCO 2005; 23:8688-8696)].
Near clinical complete response | Up to 24 weeks
  Near-cCR suggests a significant reduction in tumor size and extent, but with slight evidence of disease that stops short of the criteria for a complete clinical response, which is the total disappearance of all signs of cancer in response to treatment.
Disease free survival | Up to 3 years
  The time interval between the date of randomization and the date of the first cancer-related event, second cancer, or death from any cause, whichever occurred first.
Overall survival | Up to 3 years
  The time interval between the date of randomization to the date of death. If the patient has been alive, the time until the last follow-up is taken as the overall survival period.
Local surgery rate | Up to 24 weeks
  The local surgery rate is defined as the proportion of patients who undergo surgical intervention limited to the area of the primary tumor site, without extensive removal of surrounding tissue or organs.
Local recurrence rate | Up to 3 years
  The local recurrence rate refers to the proportion of patients in whom cancer returns at the site of the original tumor after treatment.
Distant metastasis rate | Up to 3 years
  The distant metastasis rate is defined as the proportion of patients who develop metastases at sites remote from the primary tumor location after initial treatment.
Relapse-free survival | Up to 3 years
  The time interval between the date of randomization and the date of the first cancer-related event, second cancer, or death from any cause, whichever occurred first.
Stoma-free survival | Up to 3 years
  Stoma-free survival is defined as the duration of time during which a patient with cancer, particularly colorectal or rectal cancer, remains alive without the need for a stoma following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, MD, Ph D, Study Chair — Sun Yat-sen University
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No